CLINICAL TRIAL: NCT03626727
Title: Open-label Clinical Trial to Evaluate the Efficacy of Sodium Oxybate (Xyrem®) in the Treatment of Two Under-recognized Clinical Conditions: Post-traumatic Narcolepsy and Post-traumatic Hypersomnia
Brief Title: Evaluation of the Efficacy of Sodium Oxybate (Xyrem®) in Treatment of Post-traumatic Narcolepsy and Post-traumatic Hypersomnia
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Target study population was extremely difficult to recruit and planned study budget was exceeded
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Charles Andrew Czeisler, MD, PhD, Baldino Professor of Sleep Medicine, Division Chief, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-P-002884
Record Dates: First submitted 2018-06-27; First posted 2018-08-13 (Actual); Last update posted 2021-03-04 (Actual); Status verified 2021-03

CONDITIONS: Hypersomnia; Narcolepsy; Traumatic Brain Injury
Keywords: Excessive Daytime Sleepiness; Prolonged sleep; Traumatic Brain Injury
MeSH Terms: conditions — Disorders of Excessive Somnolence; Narcolepsy; Brain Injuries, Traumatic | interventions — Sodium Oxybate

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Sodium Oxybate Oral Solution (Xyrem®) (Experimental): 4.5g of oral solution Xyrem will be given as a starting dose. This will be titrated up weekly to the final treatment dose of 9.0g. Participants will be on this final dose for 8 weeks.
  Interventions: Drug: Sodium Oxybate Oral Solution [Xyrem]

INTERVENTIONS:
Drug: Sodium Oxybate Oral Solution [Xyrem] — Xyrem will be given to participants to determine if it is effective in treating post-traumatic narcolepsy and post-traumatic hypersomnia

SUMMARY:
The study evaluates whether the use of Sodium Oxybate (Xyrem®) in TBI patients will be effective in reducing symptoms of post traumatic narcolepsy and post traumatic hypersomnia.

DETAILED DESCRIPTION:
Post-traumatic narcolepsy and post-traumatic hypersomnia are under-recognized clinical conditions in post-TBI patients.

Considering the high prevalence of hypersomnia, treatment difficulty, and sparse clinical studies for treatment of sleep problems in TBI patients, additional clinical trials need to be performed to provide more therapeutic options for patients and physicians. Sodium oxybate (Xyrem®) could be potentially one such option given its high efficacy in idiopathic narcolepsy patients.

From the results of animal research, as well as from cerebrospinal fluid (CSF) and autopsy findings from TBI patients, hypothalamic injury and hypocretin pathology seem to play a role in the pathogenesis of post-traumatic narcolepsy and hypersomnia. Despite lack of clear understanding of the exact mechanism of action of sodium oxybate in patients with idiopathic narcolepsy, the shared pathophysiology of the hypocretin system in post-traumatic hypersomnia and narcolepsy would suggest the possible efficacy of sodium oxybate (Xyrem®) on excessive daytime sleepiness (EDS) and prolonged sleep in patients with TBI.

In this Pilot Clinical Trial, we will test whether sodium oxybate (Xyrem®, approved for the treatment of improve wakefulness in adult patients with excessive sleepiness associated with narcolepsy) is effective in improving the sleep-wake symptoms, global functioning and quality of life of post-TBI patients with hypersomnia and narcolepsy.

ELIGIBILITY:
Inclusion Criteria:

* History of first-ever primary TBI 12 or more months ago;
* Mild to severe TBI (GCS 3-15);
* Either a) or b):

  1. Presence of subjective daytime sleepiness (ESS ≥ 10) lasting 3 months or more, and not present prior to the TBI;
  2. Long sleep duration (mean TST ≥ 9hours/24hrs or increased sleep need of at least 1-2 h per 24 h compared to pre-TBI), documented by actigraphy, lasting 3 months or more;
* Objectively demonstrated EDS (MSLT mean of 5 naps: SL ≤ 8min);
* Age: 18 - 64;
* Ability to read and understand consent form, complete questionnaires and daily sleep diary, and provide informed consent. The Folstein MMSE will be used to assess cognitive function.

Exclusion Criteria:

* Current neurologic deficit (weakness, dysarthria or dysphagia, aphasia or dysphasia); Participants with a score of <27 on Folstein MMSE will be excluded.
* History of neurologic or psychiatric disease prior to TBI;
* Epilepsy or history of seizure (whether related or unrelated to TBI);
* Body mass index (BMI) ≥ 32;
* Sleep apnea (Apnea Hypopnea Index, AHI > 15/h); -Chronic sleep restriction (≥ 2hour sleep extension on weekends from self- report, diary, or at least 14 days of actigraphy);
* Sleep-wake disturbance other than long sleep duration or sleepiness (DSPD, ASPD, Shift-work Sleep Disorder);
* Diagnosis of narcolepsy or other sleep disorder prior to TBI;
* Unwillingness to follow physician instructions relating to the concomitant use of alcohol and sodium oxybate during the study;
* History of or current substance abuse;
* Current regular CNS-affecting medication use;
* History of depression, suicidal thoughts, and/or post-traumatic stress disorder (PTSD);
* Current depression assessed by a structured clinical interview and Beck Depression Inventory (BDI);
* Abnormal liver function (LFT more than twice the upper limit of normal or serum bilirubin more than 1.5 times the upper limit of normal);
* Hypertension, heart failure, history of myocardial infarction, or abnormal EKG demonstrating clinically significant arrhythmia;
* Kidney disease (Serum creatinine >2.0mg/dl);
* Lung disease (COPD, ILD, asthma);
* On a low salt diet for medical reasons;
* An occupation that requires variable shift work or routine night shifts (work hours between 11pm and 6am);
* Pregnant, intention to become pregnant;
* Breast-feeding or plans to breastfeed;
* Succinic semialdehyde dehydrogenase deficiency.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2020-09 (Estimated); Primary Completion 2020-09-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Change in Subjective Daytime Sleepiness | Data collected on Day 1 (Baseline Visit) of the Intervention and at end of 1 week on the final dosage, which will be 2-5 weeks after the Baseline Visit.
  Change in subjective daytime sleepiness assessed through a daily questionnaire about frequency and duration of daytime naps, frequency of sleep attacks.
Change in Sleep Duration | Data collected on Day 1 (Baseline Visit) of the Intervention and at end of 1 week on the final dosage, which will be 2-5 weeks after the Baseline Visit.
  Change in sleep duration assessed by actigraphy-estimated total sleep time (TST).
Change in Clinical Condition | Data collected on Day 1 (Baseline Visit) of the Intervention and at end of 1 week on the final dosage, which will be 2-5 weeks after the Baseline Visit.
  Change in clinical condition as assessed by Clinical Global Impression (CGI) assessment. CGI assesses a clinician's view of a patient's global functioning before and after initiating medication. It is broken up into CGI-S (Severity) and CGI-I (Improvement). CGI-S is one question assesses how clinically ill a patient is at time of assessment. it is on a 1-7 scale with 1 being normal and 7 being among the most extremely ill patients. CGI-I looks at improvement in patients functioning once medication starts. it is also on a 1-7 scale with 1 being very much improved since initiation of treatment and 7 being very much worse.
Change in Subjective Daytime Sleepiness (ESS) | Data collected on Day 1 (Baseline Visit) of the Intervention and at end of 1 week on the final dosage, which will be 2-5 weeks after the Baseline Visit.
  Change in daytime sleepiness will be assessed through changes in Epworth Sleepiness Scale (ESS) scores. The ESS measures sleepiness of a participant. It is eight questions with a scale of 0 - 3 with 0 being no chance of dozing and 3 being high chance of dozing. The total score of eight questions is reported.

SECONDARY OUTCOMES:
Change in Nocturnal Sleep Quality (Frequency of nocturnal awakenings) | Data collected on Day 1 (Baseline Visit) of the Intervention and at end of 1 week on the final dosage, which will be 2-5 weeks after the Baseline Visit.
  Average change in nocturnal sleep quality assessed by a daily sleep questionnaire on frequency of nocturnal awakenings.
Change in Nocturnal Sleep Quality (Duration of nocturnal awakenings) | Data collected on Day 1 (Baseline Visit) of the Intervention and at end of 1 week on the final dosage, which will be 2-5 weeks after the Baseline Visit.
  Average change in nocturnal sleep quality assessed by a daily sleep questionnaire on duration of nocturnal awakenings.
Change in Nocturnal Sleep Quality (Subjective amount of sleep) | Data collected on Day 1 (Baseline Visit) of the Intervention and at end of 1 week on the final dosage, which will be 2-5 weeks after the Baseline Visit.
  Average change in nocturnal sleep quality assessed by a daily sleep questionnaire on subjective amount of sleep each night.
Change in Nocturnal Sleep Quality (Frequency of sleep walking) | Data collected on Day 1 (Baseline Visit) of the Intervention and at end of 1 week on the final dosage, which will be 2-5 weeks after the Baseline Visit.
  Average change in nocturnal sleep quality assessed by a daily sleep questionnaire on frequency of sleep walking.
Change in Nocturnal Sleep Quality (Frequency of hypnagogic hallucinations) | Data collected on Day 1 (Baseline Visit) of the Intervention and at end of 1 week on the final dosage, which will be 2-5 weeks after the Baseline Visit.
  Average change in nocturnal sleep quality assessed by a daily sleep questionnaire on frequency of hypnagogic hallucinations.
Change in Nocturnal Sleep Quality (Change in Pittsburgh Sleep Quality index) scores) | Data collected on Day 1 (Baseline Visit) of the Intervention and at end of 1 week on the final dosage, which will be 2-5 weeks after the Baseline Visit.
  Average change in nocturnal sleep quality assessed by changes in Pittsburgh Sleep Quality Index (PSQI) scores. The PSQI assesses sleep quality. It is broken down into seven components, with scales from 0 - 3 with 0 being better quality of sleep and 3 being a more poor quality of sleep. The Global PSQI score is taken from the sum of the seven component scores.
Change in Nocturnal Sleep Quality (actigraphy) | Data collected on Day 1 (Baseline Visit) of the Intervention and at end of 1 week on the final dosage, which will be 2-5 weeks after the Baseline Visit.
  Average change in nocturnal sleep quality measured by actigraphy.
Change in Global Functioning | Data collected on Day 1 (Baseline Visit) of the Intervention and at end of 1 week on the final dosage, which will be 2-5 weeks after the Baseline Visit.
  Change in global functioning evaluated by the Sheehan Disability Scale (SDS). The SDS assesses functional impairment in three subscales: in work/school, social, and family life. Each is subscale is 1-10 with 1 being no disability/impairment and 10 be extreme disability/impairment. These three subscales are added together to give the global functional impairment score which ranges from 0 being unimpaired to 30 being highly impaired.

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States